CLINICAL TRIAL: NCT04199377
Title: Retrospective Evaluation of Clinical and Functional Results and Survivorship of Total Knee Replacement and Total Hip Replacement, Both Isolated or Combined.
Acronym: ALLCCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLCCP
Record Dates: First submitted 2017-11-27; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: HIP REPLACEMENT; KNEE REPLACEMENT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hip or knee replacement (Experimental): total hip or knee replacement
  Interventions: Procedure: HIP KNEE REPLACEMENT

INTERVENTIONS:
Procedure: HIP KNEE REPLACEMENT — HIP KNEE REPLACEMENT

SUMMARY:
Retrospective evaluation of clinical and functional results and survivorship of total knee replacement and total hip replacement, both isolated or combined.

DETAILED DESCRIPTION:
Retrospective evaluation of clinical and functional results and survivorship of total knee replacement and total hip replacement, both isolated or combined.

Evaluation performed 1, 2, 5, 10 and 15 years after surgery

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Patients underwent total knee or hip replacement, both isolated or combined with other surgical procedures

Exclusion criteria

- Patients underwent other types of knee or hip replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
HARRIS HIP SCORE | 10 years
  scale range: 0-100; excellent results: 80-100
KNEE SOCIETY SCORE | 10 years
  scale range: 0-100; excellent results: 80-100
HARRIS HIP SCORE | 5 years
  scale range: 0-100; excellent results: 80-100
KNEE SOCIETY SCORE | 5 years
  scale range: 0-100; excellent results: 80-100

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No